CLINICAL TRIAL: NCT00406432
Title: A Steady-state Study to Assess the Pharmacokinetic Profile of Paroxetine After 14 Day Repeated Daily Dosing of the Controlled Release Paroxetine Tablet (25 mg) in Healthy Chinese Subjects
Brief Title: A Repeat Dose Pharmacokinetic Study Of Paroxetine CR Tablet In Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCR104075
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder
Keywords: BRL029060/Paroxetine CR; pharmacokinetics; repeat dose
MeSH Terms: conditions — Depressive Disorder

ARMS (1):
- Subjects receiving paroxetine (Experimental): Eligible subjects will receive single dose of paroxetine 25 milligrams controlled release formulation followed by wash-out period of 5 days. Subjects will receive multiple doses of paroxetine 25 milligrams for further 14 days.
  Interventions: Drug: Paroxetine Controlled Release Tablet

INTERVENTIONS:
Drug: Paroxetine Controlled Release Tablet — Eligible subjects will receive paroxetine controlled release tablet with dose of 25 milligrams.

SUMMARY:
The study was designed to assess the steady-state pharmacokinetic profile of paroxetine after 14 day repeated daily dosing of the controlled release tablet formulation (25 mg) in healthy Chinese subjects.

ELIGIBILITY:
Inclusion criteria:

* 19-45 years healthy Chinese subjects
* Body weight > 50 kg
* BMI between 19-25
* serological negative for HIV, syphilis and hepatitis B and C
* no abnormalities in ECG
* Female with negative pregnancy and male has no plan to have a child during and 3 months after the study.

Exclusion criteria:

* History of chronic physical/mental disease, current disease and concomitant medication

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05-09 (Actual); Primary Completion 2006-06-02 (Actual); Study Completion 2006-06-02 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters | Up to 21 days

SECONDARY OUTCOMES:
safety parameters(adverse events, lab test results,vital signs,electrocardiograph) | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China

REFERENCES:
- See also: Results for study PCR104075 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/PCR104075?search=study&study_ids=PCR104075#rs